CLINICAL TRIAL: NCT06218654
Title: Hemodynamic Instability of Patient With Spontaneous Subarachnoid Hemorrhage and Systemic Response to Endogenous Stress. Urinary and Serum Factors and Clinical Developments. Pilot Study Toward the Predictivity of Clinical Failure and Variation on Outcome in the Neurosurgical Patient (HISAHES)
Brief Title: Hemodynamic Instability of Patient With Spontaneous Subarachnoid Hemorrhage
Acronym: HISAHES
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6185
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-01

CONDITIONS: Subarachnoid Hemorrhage, Spontaneous; Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: biomarkers — Serum tests for specific cardiac troponin (cTPI), neuron-specific enolase (NSE), natriuretic peptides (NT-ProBNP), S100 protein (S100B), Soluble Suppressor of Tumorigenesis-2 (sST2), and soluble urokinase plasminogen activator receptor (suPAR) tests will be performed, as well as urinary tests for epinephrine and norepinephrine. On these samples, conducted according to clinical practice, additional measurements will also be taken for glial fibrillary acidic protein (GFAP) and ubiquitin carboxy-terminal hydrolase (UCH-L1) as specific study biomarkers on blood samples.
  All samples will be collected within 24 hours of admission to the Emergency Department (T0) and after 72 hours (T1). A sample at day 7 (T2) will be taken.

SUMMARY:
The goal of this observational study is to learn about the role of biomarkers in spontaneous subarachnoid hemorrhage (sSAH) as predictors of severity of clinical outcome. The test of biomarkers is based on regular blood and urinary samples. Blood levels of highly specific cardiac troponin (cTNI), natriuretic peptides (NT-ProBNP), S100 beta protein, neuron-specific enolase (NSE), glial fibrillary acidic protein (GFAP), ubiquitin carboxy-terminal hydrolase (UCH-L1), soluble Tumor Necrosis Factor Receptor-2 (sST2), and soluble urokinase plasminogen activator receptor (suPAR), as well as urinary levels of epinephrine and norepinephrine are the biomarkers explored. All adult participants with spontaneous subarachnoid hemorrhage are involved in the study.

The main questions aim to answer are:

* which of these molecules can be prognostic for patients' outcome
* which are the prognostic levels of these biomarkers to predict patients' outcome.

Participants will undergo blood and urinary samples during hospitalization at 24 hours, 72 hours and after 7 days.

DETAILED DESCRIPTION:
Spontaneous subarachnoid hemorrhage (sSAH) is one of the most severe neurological conditions. The hemodynamic instability due to endogenous catecholamine response and inflammatory patterns influences the risk of an unfavorable outcome and the development of clinical implications such as neurological and non-neurological issues. Serum levels of highly specific cardiac troponin (cTNI), natriuretic peptides (NT-ProBNP), S100 beta protein, neuron-specific enolase (NSE), glial fibrillary acidic protein (GFAP), ubiquitin carboxy-terminal hydrolase (UCH-L1), soluble Tumor Necrosis Factor Receptor-2 (sST2), and soluble urokinase plasminogen activator receptor (suPAR), as well as urinary levels of epinephrine and norepinephrine, can be measured as biomarkers in sSAH to explore the systemic response to the stress of bleeding. However, not all sSAH cases equally develop this endogenous cascade responsible for neurological and systemic events. There is no clear validation of threshold levels of endogenous factors applicable in clinical practice to define hemodynamic instability that has only a neurological or multi-organ impact post-SAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous subarachnoid hemorrhage, including those with perimesencephalic subarachnoid hemorrhage and aneurysmal subarachnoid hemorrhage.
* Adult patients.
* Confirmed presence of spontaneous subarachnoid hemorrhage through neuroimaging.
* Obtained informed consent for specific study biomarkers

Exclusion Criteria:

* Age <18 years.
* Post-traumatic subarachnoid hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (>18 years) diagnosed with spontaneous subarachnoid hemorrhage admitted at the Fondazione Policlinico Universitario Agostino Gemelli will be enrolled in the study. Bleeding will be defined as hemorrhage measured on CT using a volumetry program conducted by the Department of Radiology. For all patients, angioCT and angiography (performed if necessary for diagnosis) data will be collected from the initial diagnosis. Radiological images obtained at the time of diagnosis will be collected and anonymized
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and patients outcome | t0 at 24 hours, t1 at 72 hours, t2 at 7 days
  Assessing biomarkers as prognostic factors through logistic regression analysis, adjusted for confounding factors (gender, age, imaging, neurological and systemic complications) that may influence clinical outcomes (mRS).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Maria Della Pepa, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS; Anna Maria Auricchio, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy